CLINICAL TRIAL: NCT04681456
Title: Skin Cancer Oncology Radiation Evidence Registry
Acronym: SCORER
Status: Terminated | Type: Observational
Why Stopped: The study was stopped in order to reconfigure it as a PhaseII/III study
Sponsor: GenesisCare USA (Other)
Responsible Party: Sponsor
Other Study IDs: GCUSA-2020-03
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2020-12

CONDITIONS: Non-melanoma Skin Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: There is no medical intervention for the purposes of this Registry. — There is no medical intervention for the purposes of this Registry.

SUMMARY:
To collect and analyze long term safety and efficacy outcomes of patients undergoing radiotherapy for non-melanoma skin cancer. A target of 400 VMAT-treated sites is set which is estimated to be identified in approximately 350 participants. Participants referred for radiotherapy for the management of non-melanoma skin cancer.

DETAILED DESCRIPTION:
The Registry will collect information on key clinical indications and patient reported outcomes to assess the safety and efficacy of VMAT radiotherapy. Data that will be collected includes baseline data of demographic, relevant medical history, photographs, treatment schedule, and treatment outcomes. Data may be collected retrospectively in regard to previous relevant medical history, prior treatments and outcomes as well as prospectively, including treatment schedule and treatment outcomes of radiotherapy treatment.

The Registry aims to assess the safety and outcomes of treatment for up to 5 years. This Registry will be the first of its kind in the US and will provide a basis for a number of potential research publications. The Registry will also give insights into treatment delivery and potentially facilitate future improvements in patient care.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosed with a treatable non-melanoma skin cancer by referring medical practitioner
* Eligible to be treated using widefield (>50cm2) VMAT radiotherapy as determined by RO
* Patient has provided written informed consent.

Exclusion Criteria:

♦ Patients who do not consent to their involvement in the Registry.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited based on their potential eligibility to receive VMAT widefield radiotherapy treatment of their NMSC. The RO will assess if the condition is suitable for VMAT treatment, and if so, will discuss the Registry with the participant.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Participants will have their responses to radiotherapy after treatment of non-melanoma skin cancer measured and reported as number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 5 years
  To assess participant safety following treatment of non-melanoma skin cancers with radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Mantz, MD, Principal Investigator — GenesisCare USA
Locations (1):
- GenesisCare USA, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All other researchers belong to the same organization and could potentially have access to all data gathered.
Supporting Information: Study Protocol
Time Frame: 2021 or 2022
Access Criteria: Data will be stored on secured servers of the sponsoring organization and will be password protected with limited access.